CLINICAL TRIAL: NCT01349179
Title: Scan Evaluation at 9 Years of the Bone Acetabular Supporting Cups Without Cement (Couple Metal/Metal in Diameter 28 mm)
Brief Title: Scan Hip Evaluation
Acronym: ETOSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHU-089
Record Dates: First submitted 2011-02-22; First posted 2011-05-06 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Hip Arthroplasty
Keywords: Hip; Arthroplasty; Metal on metal; operated on 2002

INTERVENTIONS:
Device: Metal on metal hip arthroplasty operated on 2002 — The purpose of the study is to evaluate the presence of geodes acetabular and femoral with scan examination.

SUMMARY:
The couple of friction metal-polyethylene is regarded as the couple of reference in spite of the osteolysis induced by the wear of the polyethylene which remains the independent factor of long-term failure. This is all the more true as the patients are young, thus justifying the recourse to alternate couples of friction. The Metasul® couple was introduced on the French market under its current form in 1995 (year of its marking EC). The use of a couple of friction metal-metal (MM) is justified because it would be likely to improve longevity of the total arthroplasties of the active subjects by the reduction in osteolysis related to the wear of polyethylene. Various studies highlight evolutions different according to the types of fixing acetabular; favourable results of the not cemented cups contrasting with unsealings and the evolutionary edgings of the Metasul® cups cemented of or the cups "of cemented Weber type".

DETAILED DESCRIPTION:
Radiographies standards allow the follow-up of the total prostheses of hip but those underestimate the incidence and the extension of osteolyses perished-acetabular which are generally asymptomatic initially. The lack of international consensus on the definition of the parameters of interpretation of the radiological follow-up of the PTH makes difficult the comparison of the various results. The purpose of the study is to evaluate the presence of geodes acetabular and femoral with scan examination.

ELIGIBILITY:
Inclusion Criteria:

* Metal on metal hip arthroplasty operated on 2002
* Age older than 40 years

Exclusion Criteria:

* Expectant mothers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Realization of a scan nine years after the surgery of total hip arthroplasty | after nine years

SECONDARY OUTCOMES:
Clinical results preoperative Postel Merle d'Aubigné, Harris score preoperative and SF12 scores preoperative (before the hip surgery) | after nine years
Cooperating X-ray assessments and scan | after nine years
Realization of a X-ray and a scan then comparison of the results obtained | after nine years
Concentrations of cobalt: chrome and nickel in blood | after nine years
Rate of survival of the prosthesis | after nine years

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane DESCAMPS, MD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France